CLINICAL TRIAL: NCT02232945
Title: Banlangen Granules Anti-seasonal Influenza Study: a Randomized, Double Blind, Positive and Placebo Controlled，Clinical Study.
Brief Title: Banlangen Granules Anti-seasonal Influenza Study
Acronym: BLG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hutchison Whampoa Guangzhou Baiyunshan Chinese Medicine Company Limited (Industry)
Collaborators: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HWBY-001
Record Dates: First submitted 2012-11-18; First posted 2014-09-05 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Influenza
Keywords: influenza A (H1N1,H3N2); influenza B virus
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; banlangen

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): placebo of oseltamivir phosphate and placebo of Banlangen(Radix Isatidis) granules.
  Interventions: Drug: placebo of oseltamivir phosphate; Drug: placebo of Banlangen(Radix Isatidis) granules
- Banlangen granules & placebo (Experimental): Banlangen(Radix Isatidis) granules and placebo of oseltamivir phosphate
  Interventions: Drug: placebo of oseltamivir phosphate; Drug: Banlangen (Radix Isatidis) granules
- oseltamivir phosphate & placebo (Active Comparator): oseltamivir phosphate and placebo of Banlangen(Radix Isatidis) granules
  Interventions: Drug: oseltamivir phosphate; Drug: placebo of Banlangen(Radix Isatidis) granules

INTERVENTIONS:
Drug: placebo of oseltamivir phosphate
  Arms: Banlangen granules & placebo; placebo
Drug: oseltamivir phosphate
  Arms: oseltamivir phosphate & placebo
Drug: Banlangen (Radix Isatidis) granules
  Arms: Banlangen granules & placebo
Drug: placebo of Banlangen(Radix Isatidis) granules
  Arms: oseltamivir phosphate & placebo; placebo

SUMMARY:
This study aimed to evaluate the efficacy and safety of the nature herbal medicine Banlangen granules in patients infected with seasonal influenza A (H1N1,H3N2) and influenza B virus.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Patients have confirmed influenza A(H1N1,H3N2) or influenza B virus infection by real time PCR
2. age between 18-65 years old
3. axillary temperature ≥38ºC and with at least two constitutional symptoms (headache, chill, myalgia ，or fatigue) and one respiratory symptom (cough ，sore throat,or coryza) .
4. Illness onset had to be within 36 hours, and informed consent was obtained.

Exclusion criteria:

1. age younger than 18 or older than 65 years old.
2. patients confirmed with bronchitis, pneumonia,pleural effusion and interstitial lung disease by Chest imaging (chest X-ray or CT) .
3. Blood routine screening tests shows numeration of leukocyte 10.0×109/L or Neutrophil percentage ≥80%.
4. Those have got suppurative tonsillitis or cough purulent sputum.
5. Those with underling primary disorders, such as hematological disease, chronic obstructive pulmonary disease（FEV1/FVC<70％，FEV1/ predicated value<50％； or respiratory failure or right heart failure）， hepatic disease（ALT or AST≥triple ULN）, renal disease（Serum Creatinine>2mg/dL）,chronic congestive heart failure( NYHA Ⅲ-IV)

7. Patient is allergic to the study medication(s). 8. Women who are pregnant or may possibly become pregnant or are lactating with a positive urine pregnant test, obesity (abody mass index (BMI) of 25 kg/m2 or more).

9. Those with immunodeficiency ,such as malignant tumor ; Organs or bone marrow transplantation ; AIDS ;or taking immune inhibitors during the last 3 months.

10. Doubt or does alcohol/drug abuse of history. 11. Those have participated in other clinical trial within three month before study randomization.

12. Two weeks before the test , those with acute respiratory Infection，otitis,or nasosinusitis .

13. Those already vaccinated or who will receive influenza vaccine. 14. other reasons not suitable for enrollment based on the investigator's discretion.

The primary efficacy endpoint:

1. The primary end point was the duration of illness which was defined as the time from onset of symptoms to the alleviation of the ten influenza-like symptoms including , nasal obstruction, running nose, cough, sore throat, headache, fatigue, myalgia, chills and sweating.
2. The time to defervescence, defined as the time from the first dose of study medication to the time when the body temperature declined to lower than 37.4ºC and was sustained for at least 24 hours.

Secondary efficacy endpoint:

The secondary end points included: 1) viral shedding duration, defined as the time from the illness onset to the first time the viral nucleic acid test was negative; 2) the severity of the disease,assessed by an area under the curve (AUC) analysis of a total of nine influenza-like symptom scores, the AUC was calculated as the product of the daily symptom scores times the duration of illness;3)frequency of Usage of Acetaminophen;4)and incidence of secondary complications of influenza, such as otitis, bronchitis, pneumonia，Nasosinusitis ,suppurative tonsillitis,acute parotitis，Reye'ssyndrome，central nervous system disease, Myocarditis and pericarditis, acute myositis, and toxic shock syndrome.5) economic evaluation.

Specimen:

the pharyngeal or the throat swab，blood. Pharyngea /throat secretions will be obtained from the upper respiratory tract of each patient.

All specimens will be stored at -80℃ in virus laboratory of the first affiliated hospital of guangzhou medical university for 5 years.

ELIGIBILITY:
Inclusion Criteria:

with confirmed influenza A(H1N1,H3N2) or influenza B virus infection by real time RT-PCR (rRT-PCR), age between 18-65 years old, axillary temperature ≥38ºC and with at least two constitutional symptoms (headache, chill, myalgia ，or fatigue) and one respiratory symptom (cough ，sore throat,or coryza) . Illness onset had to be within 36 hours, and informed consent was obtained.

Exclusion Criteria:

1. age younger than 18 or older than 65 years old.
2. patients confirmed with bronchitis, pneumonia,pleural effusion and interstitial lung disease by Chest imaging (chest X-ray or CT) .
3. Blood routine screening tests shows numeration of leukocyte 10.0×109/L or Neutrophil percentage ≥80%.
4. Those have got suppurative tonsillitis or cough purulent sputum.
5. Those with underling primary disorders, such as hematological disease, chronic obstructive pulmonary disease（FEV1/FVC<70％，FEV1/ predicated value<50％； or respiratory failure or right heart failure）， hepatic disease（ALT or AST≥triple ULN）, renal disease（Serum Creatinine>2mg/dL）,chronic congestive heart failure( NYHA Ⅲ-IV)

7. Patient is allergic to the study medication(s). 8. Women who are pregnant or may possibly become pregnant or are lactating with a positive urine pregnant test, obesity (abody mass index (BMI) of 25 kg/m2 or more).

9. Those with immunodeficiency ,such as malignant tumor ; Organs or bone marrow transplantation ; AIDS ;or taking immune inhibitors during the last 3 months.

10. Doubt or does alcohol/drug abuse of history. 11. Those have participated in other clinical trial within three month before study randomization.

12. Two weeks before the test , those with acute respiratory Infection，otitis,or nasosinusitis .

13. Those already vaccinated or who will receive influenza vaccine. 14.other reasons not suitable for enrollment based on the investigator's discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Improving the flu-like symptoms, such as fever etc | 21+7days
  The primary end point was the duration of illness which was defined as the time from onset of symptoms to the alleviation of the ten influenza-like symptoms including , nasal obstruction, running nose, cough, sore throat, headache, fatigue, myalgia, chills and sweating.
Improving the flu-like symptoms, such as fever etc | 21+7days
  The time to defervescence, defined as the time from the first dose of study medication to the time when the body temperature declined to lower than 37.4ºC and was sustained for at least 24 hours.

SECONDARY OUTCOMES:
others | 21+7days
  viral shedding duration, defined as the time from the illness onset to the first time the viral nucleic acid test was negative
Others | 21+7days
  the severity of the disease,assessed by an area under the curve (AUC) analysis of a total of nine influenza-like symptom scores, the AUC was calculated as the product of the daily symptom scores times the duration of illness
Others | 21+7days
  frequency of Usage of Acetaminophen
Others | 21+7days
  incidence of secondary complications of influenza
Others | 21+7days
  economic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan Zhong, PhD, Study Chair — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li ZT, Li L, Chen TT, Li CY, Wang DQ, Yang ZF, Zhong NS. Efficacy and safety of Ban-Lan-Gen granules in the treatment of seasonal influenza: study protocol for a randomized controlled trial. Trials. 2015 Mar 28;16:126. doi: 10.1186/s13063-015-0645-x. PMID 25873046